CLINICAL TRIAL: NCT05581095
Title: EMBRACE MOMS 2 BE: A Pilot Feasibility, Acceptability, and Preliminary Efficacy Study of a Mindful Eating Self-Help Program for Women Who Binge Eat During Pregnancy
Brief Title: Empowering Mindfulness, Body Respect, and Compassionate Eating Among Women Who Binge Eat During Pregnancy
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: We have experienced difficulty with recruitment and will be altering the study's eligibility criteria.
Sponsor: University of North Carolina, Charlotte (Other)
Responsible Party: Principal Investigator, Jennifer B. Webb, Ph.D., Associate Professor, University of North Carolina, Charlotte
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRBIS-19-0680
Record Dates: First submitted 2022-07-16; First posted 2022-10-14 (Actual); Last update posted 2023-05-23 (Actual); Status verified 2023-05

CONDITIONS: Pregnancy; Binge Eating
MeSH Terms: conditions — Bulimia

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial of mindful eating self-help book (group 1) vs. mindful eating self-help book + companion smartphone app (group 2)
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindful Eating Self-Help Book Only (Active Comparator): Participants will be invited to read about and practice a variety of mindful eating-related strategies over the course of 10 weeks based on Dr. Michelle May & Dr. Kari Anderson's self-help book entitled, "Eat What You Love, Love What You Eat for Binge Eating". Participants will also be asked to complete a weekly electronic log describing their experiences with the weekly mindfulness-based practices.
  Interventions: Behavioral: Mindful Eating Self-Help Program
- Mindful Eating Self-Help Book + Smartphone App (Experimental): Participants will be invited to read about and practice a variety of mindful eating-related strategies over the course of 10 weeks based on Dr. Michelle May & Dr. Kari Anderson's self-help book entitled, "Eat What You Love, Love What You Eat for Binge Eating". In addition, participants will be asked to use the companion Am I Hungry? Mindful Eating Virtual Coach smartphone application three times daily. Participants will also be asked to complete a weekly electronic log describing their experiences with the weekly mindfulness-based practices.
  Interventions: Behavioral: Mindful Eating Self-Help Program; Behavioral: Mindful Eating Smartphone Application (Am I Hungry? Virtual Coach)

INTERVENTIONS:
Behavioral: Mindful Eating Self-Help Program — 10-week exposure to mindful eating principles and practices outlined in the Eat What You Love, Love What You Eat for Binge Eating book
Behavioral: Mindful Eating Smartphone Application (Am I Hungry? Virtual Coach) — 10-week exposure to using a mindful eating mobile phone application daily.
  Arms: Mindful Eating Self-Help Book + Smartphone App

SUMMARY:
Primary Study Aims:

1. To evaluate the feasibility, acceptability, and preliminary efficacy of a 10-week mindful eating self-help program for women who binge eat during pregnancy. Primary efficacy targets will include measures of mindful eating and binge eating. Secondary efficacy targets will involve measures of body image and well-being.
2. To evaluate the incremental utility of adding use of a companion mindful eating smart phone application for enhancing the acceptability and preliminary efficacy of the program.
3. To gain insights into ways in which this program may be better tailored to the experiences of pregnancy for future program adaptation and refinement.

DETAILED DESCRIPTION:
Research suggests that binge eating during pregnancy may adversely impact maternal-child health and well-being. For example, clinical evidence cites binge eating as a risk factor for increased gestational weight gain, cesarean delivery, giving birth to infants who are large for gestational age (LGA), and is associated with additional maternal susceptibility for cardiometabolic dysregulation and its complications at this critical maturational period . Nevertheless, surprisingly despite the growth in epidemiological investigations of eating disorders during pregnancy, no studies to date have specifically evaluated a behavioral intervention during pregnancy to address binge eating concerns within this population. Therefore, there is significant need to address this gap in order to develop, evaluate, and disseminate evidence-based behavioral interventions for women struggling with binge eating during pregnancy. One growing area of scholarship is implementing self-help approaches as a means of increasing availability to evidence-based behavioral health interventions for individuals who may not otherwise be able to access these treatments. At the same time, interventions that incorporate mindful eating have recently shown promise as an effective intervention for reducing binge eating and overeating in a wide range of clinical and community samples. These interventions most often conducted over a period ranging between 6-20 weeks of varying formats (e.g., group, in-person versus combination with remote support, etc.), and intensities (e.g., weekly versus bi-weekly, etc.), typically introduce participants to the concepts of mindfulness, provide opportunities to engage in mindfulness meditation practices, apply mindfulness skills to the process of eating via eating-related meditations and other similar exercises including appetite awareness training and encourage between-session home practice. The Am I Hungry? Mindful Eating Program for Binge Eating was used as a model for the present study. In the original pilot investigation a sample of women with binge eating disorder engaged in a 10-week group mindful eating-based treatment program. Results indicated significant reductions in binge eating severity and psychological distress by the final assessment period which were sustained at 1-year follow-up. We have adapted this approach in order to evaluate it in a guided self-help format with and without access to a companion smartphone application and among other things to directly assess not only changes in binge eating but also those related to more adaptive eating processes such as mindful and intuitive eating styles.

ELIGIBILITY:
Inclusion Criteria:

* female (assigned sex at birth)
* able to read and write in English
* between the ages of 18-40
* lives in the United States
* between 13-16 weeks pregnant (gestation) with a singleton
* owns an iPhone or iPad
* reports engaging in recurrent binge eating (i.e., reporting engaging in at least 1 binge eating episode per week for the last 28 days according to the EDE-Qi)
* has access to a computer or tablet with Internet
* being regularly followed by a healthcare provider during their pregnancy

Exclusion Criteria:

* reports current smoking or substance abuse
* reports elevated depression (i.e., a score of 13 or higher on the EPDS)
* reports current suicidal ideation (assessed on the EPDS)
* reports anorexia, purging or compensatory behavior (both assessed on the EDE-Qi)
* reports a history of being hospitalized for mental health treatment in the last 6 months
* reports use of medications that are taken to affect appetite or metabolism (e.g., insulin)
* is currently in therapy for treating binge eating
* reports serious cardiovascular morbidity (e.g., hypertension)
* reports uncontrolled or untreated thyroid disease
* reports a history of 3 or more miscarriages, weakened cervix, or persistent bleeding during the first 12 weeks of pregnancy
* reports being unable to commit to participate fully in the 10-week program (i.e., read from the self-help book weekly, utilize the smartphone application daily, submit weekly logs of their experiences)
* individuals seeking a dieting approach to weight management during pregnancy

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-08 (Estimated); Primary Completion 2024-06 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Enrollment | 6 months after opening enrollment
  percent enrollment within 6 months of opening recruitment
Attrition | throughout the 10-week program
  percent of participants who dropped out
Program Satisfaction | after week 10
  participant satisfaction questionnaire
App Usability | after week 10
  app usability questionnaire
Mindful Eating | baseline, after week 5 (midpoint), after week 10 (immediate post)
  Mindful Eating Inventory (MEI)
Binge Eating | baseline, after week 5 (midpoint), after week 10 (immediate post)
  Eating Disorders Examination-Questionnaire with Instructions (EDE-Qi)
Intuitive Eating | baseline, after week 5 (midpoint), after week 10 (immediate post)
  Intuitive Eating Scale-2 (IES-2)

SECONDARY OUTCOMES:
Body Image | baseline, after week 5 (midpoint), after week 10 (post-program)
  Body Image in Pregnancy Scale (BIPS)
General Well-being | baseline, after week 5 (midpoint), after week 10 (post-program)
  General Well-being: Warwick-Edinburgh Mental Well-being Scale (WEMWBS)
COVID-19-related Well-being | baseline, after week 5 (midpoint), after week 10 (post-program)
  Perinatal COVID-19-related Well-being (COPE-IU)
Mindful Self-Care | baseline, after week 5 (midpoint), after week 10 (immediate post)
  Mindful Self-Care Scale (MSCS)
Weight Bias Internalization | baseline, after week 5 (midpoint), after week 10 (immediate post)
  Weight Bias Internalization Scale-Modified (WBIS-M)
Physical Activity | baseline, after week 5 (midpoint), after week 10 (immediate post)
  International Physical Activity Questionnaire-Short Form (IPAQ-SF)
Depression | baseline, after week 5 (midpoint), after week 10 (immediate post)
  Edinburgh Postnatal Depression Scale (EPDS)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer B Webb, PhD, Principal Investigator — UNC Charlotte; V Gil-Rivas, PhD, Principal Investigator — UNC Charlotte
Locations (1):
- UNC Charlotte, Charlotte, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No